CLINICAL TRIAL: NCT01740479
Title: Randomized Comparative Effectiveness Study of Complete vs Culprit-only Revascularization Strategies to Treat Multi-vessel Disease After Early Percutaneous Coronary Intervention (PCI) for ST-segment Elevation Myocardial (STEMI) Infarction
Brief Title: Complete vs Culprit-only Revascularization to Treat Multi-vessel Disease After Early PCI for STEMI
Acronym: COMPLETE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: COMPLETE-2012
Record Dates: First submitted 2012-11-27; First posted 2012-12-04 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Acute Myocardial Infarction; Coronary Artery Disease
Keywords: STEMI; ticagrelor; multi-vessel disease; culprit lesion
MeSH Terms: conditions — Coronary Artery Disease; ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complete Revascularization Strategy (Active Comparator): Complete Revascularization Strategy (Staged Non-Culprit Lesion PCI plus Optimal Medical Therapy): Staged PCI using second generation drug eluting stents (Promus Element Plus drug-eluting stent or newer version in this series is strongly recommended) of all suitable non-culprit lesions.
  All patients, regardless of randomized treatment allocation will receive optimal medical therapy consisting of risk factor modification and use of evidence-based therapies (including low dose acetylsalicylic acid (ASA) and ticagrelor).
  Interventions: Procedure: Complete Revascularization Strategy
- Optimal Medical Therapy Alone (No Intervention): Culprit lesion only Revascularization Strategy (Optimal Medical Therapy Alone): No further revascularization of non-culprit lesions.
  All patients, regardless of randomized treatment allocation will receive optimal medical therapy consisting of risk factor modification and use of evidence-based therapies (including low dose ASA and ticagrelor).

INTERVENTIONS:
Procedure: Complete Revascularization Strategy — Staged PCI using second generation drug eluting stents (Promus Element Plus drug-eluting stent or newer version in this series is strongly recommended) of all suitable non-culprit lesions plus optimal medical therapy.
  Other Names: Staged Non-Culprit Lesion PCI plus Optimal Medical Therapy
  Arms: Complete Revascularization Strategy

SUMMARY:
To determine whether, on a background of optimal medical therapy, including ticagrelor, opening of all suitable narrowings or blockages found at the time of primary PCI for an acute heart attack is better than treating only the culprit lesion in patients with multi-vessel disease.

DETAILED DESCRIPTION:
To determine if a strategy of multivessel revascularization involving PCI of all suitable non-infarct related artery lesions plus optimal medical therapy is superior to a strategy of optimal medical therapy alone in reducing (1) the composite outcome of cardiovascular (CV) death or new myocardial infarction (MI), or (2) the composite of CV death, new MI or ischemia driven revascularization (IDR) in patients with multivessel disease who have undergone early successful culprit lesion PCI for STEMI.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women within 72 hours after successful PCI (preferably using a drug eluting stent) to the culprit lesion for STEMI. PCI for STEMI can be either primary PCI or rescue PCI for failed fibrinolysis or a combination strategy where PCI is performed routinely 3-12 hours after fibrinolysis AND
2. Multi-vessel disease defined as at least 1 additional non-infarct related coronary artery lesion that is at least 2.5 mm in diameter that has not been stented as part of the primary PCI and that is amenable to successful treatment with PCI and has:

   * At least 70% diameter stenosis (visual estimation) or
   * At least 50% diameter stenosis (visual estimation) with fractional flow reserve (FFR) ≤ 0.80

Exclusion Criteria:

1. Planned revascularization of non-culprit lesion
2. Planned surgical revascularization
3. Non-cardiovascular co-morbidity reducing life expectancy to < 5 years
4. Any factor precluding 5 year follow-up
5. Prior Coronary Artery Bypass Graft (CABG) Surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4042 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
Composite of Cardiovascular death or new myocardial Infarction | over duration of follow-up (average of approximately 4 years)
  Co-primary outcome: CV death or new MI
Composite of cardiovascular death, new myocardial infarction or ischemia-driven revascularization | over duration of follow-up (average of approximately 4 years)
  Co-primary outcome: CV death, new MI or IDR

SECONDARY OUTCOMES:
Composite of CV death, new MI, ischemia-driven revascularization or hospitalization for unstable angina or heart failure | Over duration of follow-up (average of approximately 4 years)

OTHER OUTCOMES:
Major Bleeding | Over duration of follow-up (average of approximately 4 years)

CONTACTS AND LOCATIONS:
Overall Officials: Shamir R Mehta, MD, MSc, Principal Investigator — McMaster University
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dehghani P, Cantor WJ, Wang J, Wood DA, Storey RF, Mehran R, Bainey KR, Welsh RC, Rodes-Cabau J, Rao S, Lavi S, Velianou JL, Natarajan MK, Ziakas A, Guiducci V, Fernandez-Aviles F, Cairns JA, Mehta SR. Complete Revascularization in Patients Undergoing a Pharmacoinvasive Strategy for ST-Segment-Elevation Myocardial Infarction: Insights From the COMPLETE Trial. Circ Cardiovasc Interv. 2021 Aug;14(8):e010458. doi: 10.1161/CIRCINTERVENTIONS.120.010458. Epub 2021 Jul 29. PMID 34320839
- [Derived] Pinilla-Echeverri N, Mehta SR, Wang J, Lavi S, Schampaert E, Cantor WJ, Bainey KR, Welsh RC, Kassam S, Mehran R, Storey RF, Nguyen H, Meeks B, Wood DA, Cairns JA, Sheth T. Nonculprit Lesion Plaque Morphology in Patients With ST-Segment-Elevation Myocardial Infarction: Results From the COMPLETE Trial Optical Coherence Tomography Substudys. Circ Cardiovasc Interv. 2020 Jul;13(7):e008768. doi: 10.1161/CIRCINTERVENTIONS.119.008768. Epub 2020 Jul 10. PMID 32646305
- [Derived] Mehta SR, Wood DA, Storey RF, Mehran R, Bainey KR, Nguyen H, Meeks B, Di Pasquale G, Lopez-Sendon J, Faxon DP, Mauri L, Rao SV, Feldman L, Steg PG, Avezum A, Sheth T, Pinilla-Echeverri N, Moreno R, Campo G, Wrigley B, Kedev S, Sutton A, Oliver R, Rodes-Cabau J, Stankovic G, Welsh R, Lavi S, Cantor WJ, Wang J, Nakamya J, Bangdiwala SI, Cairns JA; COMPLETE Trial Steering Committee and Investigators. Complete Revascularization with Multivessel PCI for Myocardial Infarction. N Engl J Med. 2019 Oct 10;381(15):1411-1421. doi: 10.1056/NEJMoa1907775. Epub 2019 Sep 1. PMID 31475795
- [Derived] Mehta SR, Wood DA, Meeks B, Storey RF, Mehran R, Bainey KR, Nguyen H, Bangdiwala SI, Cairns JA; COMPLETE Trial Steering Committee and Investigators. Design and rationale of the COMPLETE trial: A randomized, comparative effectiveness study of complete versus culprit-only percutaneous coronary intervention to treat multivessel coronary artery disease in patients presenting with ST-segment elevation myocardial infarction. Am Heart J. 2019 Sep;215:157-166. doi: 10.1016/j.ahj.2019.06.006. Epub 2019 Jun 18. PMID 31326681